CLINICAL TRIAL: NCT02873988
Title: Regeneration of Bronchial Epithelium During Chronic Obstructive Pulmonary Disease
Acronym: EPITHREGENCOPD
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA11017
Record Dates: First submitted 2016-08-10; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- patients with COPD: patients with COPD
  Interventions: Other: bronchial epithelial cell culture
- patients without COPD: patients without COPD
  Interventions: Other: bronchial epithelial cell culture

INTERVENTIONS:
Other: bronchial epithelial cell culture

SUMMARY:
Airway epithelium integrity is essential to maintain its role of mechanical and functional barrier. Recurrent epithelial injuries require a complex mechanism of repair to restore its integrity. In chronic obstructive pulmonary disease (COPD), an abnormal airway epithelial repair may participate in airway remodelling. The objective was to determine if airway epithelial wound repair of airway epithelium is abnormal in COPD.

DETAILED DESCRIPTION:
Patients scheduled for lung resection were prospectively recruited. Demographic, clinical data and pulmonary function tests results were recorded. Emphysema was visually scored and histological remodelling features were noted. Primary bronchial epithelial cells (BEC) were extracted and cultured for wound closure assay. The investigators determined the mean speed of wound closure (MSWC) and cell proliferation index, matrix metalloprotease (MMP)-2, MMP-9 and cytokines levels in supernatants of BEC 18 hours after cell wounding. In a subset of patients, bronchiolar epithelial cells were also cultured for wound closure assay for MSWC analyze.

ELIGIBILITY:
Inclusion Criteria:

6 Patients scheduled for lung resection for cancer

Exclusion Criteria:

* Patients with asthma, cystic fibrosis, bronchiectasis or pulmonary fibrosis were excluded

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for lung resection for cancer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean speed of wound closure (MSWC) of wounded bronchial epithelial cell culture obtained from COPD and control patients | hour 18

SECONDARY OUTCOMES:
Cell proliferation index in supernatants of bronchial epithelial cells 18 hours after cell wounding. | hour 18
Matrix metalloprotease (MMP)-2 level in supernatants of bronchial epithelial cells 18 hours after cell wounding. | hour 18
Matrix metalloprotease (MMP)-9 level in supernatants of bronchial epithelial cells 18 hours after cell wounding. | hour 18
Cytokines levels in supernatants of bronchial epithelial cells 18 hours after cell wounding. | hour 18

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Perotin JM, Adam D, Vella-Boucaud J, Delepine G, Sandu S, Jonvel AC, Prevost A, Berthiot G, Pison C, Lebargy F, Birembaut P, Coraux C, Deslee G. Delay of airway epithelial wound repair in COPD is associated with airflow obstruction severity. Respir Res. 2014 Nov 27;15(1):151. doi: 10.1186/s12931-014-0151-9. PMID 25427655